CLINICAL TRIAL: NCT02365064
Title: PAP to PAP: CPAP vs ASV for Insomnia Randomized Controlled Trial
Brief Title: CPAP vs ASV for Insomnia
Acronym: P2P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 682031-1_MA20150206
Record Dates: First submitted 2015-02-10; First posted 2015-02-18 (Estimated); Results first posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-05

CONDITIONS: Insomnia; Sleep-Disordered Breathing
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Positive Airway Pressure (Active Comparator): Continuous positive airway pressure (CPAP) intervention as active comparator. Provides a fixed pressure for both inspiration and expiration.
  Interventions: Device: AirCurve 10 ASV
- Adaptive Servo-Ventilation (Experimental): Adaptive servo-ventilation (ASV) positive airway pressure as experimental intervention. Provides a higher pressure for inspiration and a lower pressure for expiration with changes in the pressure support level to meet a target minute ventilation.
  Interventions: Device: AirCurve 10 ASV

INTERVENTIONS:
Device: AirCurve 10 ASV — Device is able to provide both ASV therapy and CPAP therapy modes.
  Other Names: VPAP Adapt, AutoSet CS2

SUMMARY:
The study will determine which of two different types of positive airway pressure (PAP therapy) modes are more effective in reducing sleep breathing events in chronic insomnia patients and in decreasing insomnia severity.

DETAILED DESCRIPTION:
Patients presenting to the sleep clinic with a primary complaint of insomnia will be potential participants for this study. Following diagnostic polysomnography (PSG) testing, insomnia patients diagnosed with SDB and meeting inclusion criteria will be randomized to a PAP treatment arm, CPAP or ASV. Participants will complete titration studies with their assigned PAP mode and attend clinical follow-up appointments over a 14-16 week timeframe. Titration PSG studies will assess PAP pressure needs to ensure that patients are receiving optimal therapy at all times during this study. PAP adaptation barriers will be addressed as they arise during the study, because it is important that participants are able to use PAP therapy nightly during participation in this protocol. Baseline scores on insomnia severity, sleep quality, subjective insomnia parameters, sleep related impairment, and quality of life will be compared to outcome measures at the 4 month mark. Pre-treatment and post-treatment objective improvements on sleep studies will also be compared including sleep breathing indices, sleep consolidation indices, and objective data download information.

ELIGIBILITY:
Inclusion Criteria:

* Primary complaint of insomnia when presenting at clinic
* Diagnosis of moderate to severe insomnia through the Insomnia Severity Index (ISI) with a score ≥ 15
* Meet diagnostic criteria of Insomnia Disorder (per American Academy of Sleep Medicine)
* Diagnosis of SDB, either OSA as determined by an AHI ≥ 5 events/hour or UARS with a RDI ≥ 15 events/hour and AHI < 5 events/hour
* Naïve to treatment for sleep-disordered breathing (SDB), including CPAP, APAP, ASV; mandibular repositioning devices (MRDs), and any other nasal or oral therapy with a primary indication of treating SDB
* Able to fully understand study information in English and sign informed consent

Exclusion Criteria:

* Primary complaint of sleep-disordered breathing or issues with apneas during sleep
* Severe respiratory disorder or severe sleep disorder such as restless leg syndrome (RLS), idiopathic hypersomnia, or narcolepsy
* BMI > 30 kg/m2
* Epworth Sleepiness Scale (ESS) score ≥ 10
* Frequent napping behavior, such as a few times a week or more
* Anticipated changes to start or stop sedative or psychotropic medications during the course of the trial
* Medical history of congestive heart failure (CHF) or other potentially unstable cardiac disease as well as chronic lung diseases or other debilitating medical conditions that manifest as more prominent in the patient's health compared to their sleep complaints
* Daily use of opiate medications
* Known contraindications to PAP therapy as listed in the indication for use
* Requires a CPAP (fixed) pressure > 20 cm H2O
* Inability to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry Krakow, MD, Principal Investigator — Sleep & Human Health Institute
Locations (1):
- Maimonides Sleep Arts & Sciences, Albuquerque, New Mexico, United States

REFERENCES:
- [Derived] Krakow B, McIver ND, Ulibarri VA, Krakow J, Schrader RM. Prospective Randomized Controlled Trial on the Efficacy of Continuous Positive Airway Pressure and Adaptive Servo-Ventilation in the Treatment of Chronic Complex Insomnia. EClinicalMedicine. 2019 Aug 8;13:57-73. doi: 10.1016/j.eclinm.2019.06.011. eCollection 2019 Aug. PMID 31517263

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Continuous Positive Airway Pressure | Adaptive Servo-Ventilation
Started | 31 | 47
Included in ITT Analysis | 29 | 32
Completed | 21 | 19
Not Completed | 10 | 28
Not completed — Patients met baseline exclusion requirem | 2 | 15
Not completed — Withdrawal by Subject | 6 | 9
Not completed — Treatment intolerance | 2 | 4

BASELINE CHARACTERISTICS:
Population: Baseline information available for ITT
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Positive Airway Pressure | Adaptive Servo-Ventilation | Total
Number analyzed (Participants) | 29 | 32 | 61
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 44.95 [39.14 to 50.76] | 45.89 [40.26 to 51.52] | 45.44 [41.51 to 49.37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 23 | 42
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 8 | 13
  Not Hispanic or Latino | 24 | 24 | 48
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity Index
Description: Change in insomnia severity from baseline to 4 months as measured by subjective questionnaire. The Insomnia Severity Index has seven questions. The seven answers are added up for a total score. Scores range from 0 - 28. A higher score indicates a more severe degree of insomnia.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuous Positive Airway Pressure | Adaptive Servo-Ventilation
Number analyzed (Participants) | 21 | 19
units on a scale | 9.29 (6.57) | 13.21 (5.17)

2. Secondary Outcome: Sleep Quality Rating
Description: 8 point Likert scale for change in subjective sleep quality from baseline to 4 months. Lower scores indicated more positive sleep quality. A score 0 indicates excellent sleep quality, and a score of 7 indicates very poor sleep quality
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Continuous Positive Airway Pressure | Adaptive Servo-Ventilation
Number analyzed (Participants) | 21 | 19
score on a scale | 1.06 (1.00) | 1.65 (1.13)

3. Secondary Outcome: Global Morning Rating
Description: Change in subjective rating from baseline to 4 months based on a 0-100% scale. Lower scores equal a more positive experience
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuous Positive Airway Pressure | Adaptive Servo-Ventilation
Number analyzed (Participants) | 21 | 19
units on a scale | 15.39 (20.03) | 24.33 (13.15)

4. Secondary Outcome: Sleep Onset Latency
Description: Change in from baseline to 4 months in sleep onset time (minutes)
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Continuous Positive Airway Pressure | Adaptive Servo-Ventilation
Number analyzed (Participants) | 21 | 19
minutes | -6.09 (44.39) | 7.17 (26.90)

5. Secondary Outcome: Wake After Sleep Onset (WASO)
Description: Change from baseline to 4 months for WASO in minutes
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Continuous Positive Airway Pressure | Adaptive Servo-Ventilation
Number analyzed (Participants) | 21 | 19
minutes | 5.72 (58.73) | -0.12 (61.88)

6. Secondary Outcome: Sleep Efficiency
Description: Change from baseline to 4 months in sleep efficiency (total sleep time/time in bed)
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: percentage of time in bed
Arm/Group | Continuous Positive Airway Pressure | Adaptive Servo-Ventilation
Number analyzed (Participants) | 21 | 19
percentage of time in bed | 0.75 (16.68) | -2.85 (16.05)

ADVERSE EVENTS:
Time Frame: 4 months
Description: Participants were asked to report side effects commonly related to CPAP usage, including:
  Drying of the nose, mouth or throat, Nosebleed, Ear or sinus discomfort, Eye irritation, Skin rashes Participants may report multiple side effects
Arm/Group | Continuous Positive Airway Pressure | Adaptive Servo-Ventilation
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 20/21 | 16/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Continuous Positive Airway Pressure (N=21) | Adaptive Servo-Ventilation (N=19)
mask leak (Respiratory, thoracic and mediastinal disorders) | 20 | 16 — Mask leak is a common side effect to CPAP treatment, and can lead to dry mouth (from mask/ mouth leak), congestion, and eye irritation
dry mouth (Respiratory, thoracic and mediastinal disorders) | 19 | 16 — Dry mouth is a common complaint usually caused by mask leak or mouth breathing while using PAP
skin irritation (Skin and subcutaneous tissue disorders) | 15 | 13 — Skin irritation due to wearing a mask at night
mask related insomnia (Respiratory, thoracic and mediastinal disorders) | 13 | 11 — Difficulty sleeping due to wearing a CPAP mask
mouth leak (Respiratory, thoracic and mediastinal disorders) | 12 | 11 — Discomfort due to air leaking from the mouth during CPAP use
congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 12 — Nasal congestion due to CPAP use
skin crease from mask (Skin and subcutaneous tissue disorders) | 12 | 9 — Facial marks due to wearing a CPAP mask at night
nose tickle/ burn (Respiratory, thoracic and mediastinal disorders) | 11 | 9 — Discomfort in nasal passages while using CPAP
aerophagia (Respiratory, thoracic and mediastinal disorders) | 9 | 7 — Discomfort from swallowing air during CPAP use
eye irritation (Respiratory, thoracic and mediastinal disorders) | 7 | 8 — Eye irritation due to mask leak (air leaking into eyes) during CPAP use

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-07): https://cdn.clinicaltrials.gov/large-docs/64/NCT02365064/Prot_SAP_000.pdf